CLINICAL TRIAL: NCT06073509
Title: Watch Your HeaRT Study - Screening and Risk Analysis of Atrial Fibrillation and Other Cardiac Arrhythmias and Diseases After Radiotherapy for Breast Cancer
Brief Title: Atrial Fibrillation and Other Cardiac Arrhythmias and Diseases After Radiotherapy for Breast Cancer : Watch Your HeaRT
Acronym: WATCH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sophie JACOB (Other Government)
Collaborators: Clinique Pasteur Toulouse (Other); Centre Francois Baclesse (Other); Institut Curie (Other)
Responsible Party: Sponsor-Investigator, Sophie JACOB, Study Coordinator, Institut de Radioprotection et de Surete Nucleaire
Organization: Institut de Radioprotection et de Surete Nucleaire (Other Government)
Other Study IDs: WATCH_2023
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Radiation Toxicity; Atrial Fibrillation; Cardiac Arrhythmia; Cardiac Disease
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries; Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases | interventions — Mass Screening; Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients treated with RT 5 years ago: Retrospective and cross-sectional data collection based on a medical questionnaire and screening for atrial fibrillation and other cardiac arrhythmias and diseases.
  Interventions: Diagnostic Test: Screening for atrial fibrillation and other cardiac arrhythmias and diseases

INTERVENTIONS:
Diagnostic Test: Screening for atrial fibrillation and other cardiac arrhythmias and diseases — In addition to retrospective data collection based on a medical questionnaire, a 5-year post-RT cardiovascular screening will include:
  * connected smartwatches for atrial fibrillation screening
  * complete ECG for other cardiac arrhythmias
  * echocardiography for other cardiac diseases (including cardiac dysfunction, cardiomyopathy, valvulopathy, ...)

SUMMARY:
The goal of this interventional study is to evaluate the risk of atrial fibrillation (AF) and other cardiac arrhythmias and diseases in breast cancer patients treated with radiation therapy (RT).

In addition to regular follow-up of patients by the radiation oncologist for 5 years, cardiovascular screening at the end of follow-up, combining the use of a connected watch and a cardiological check-up, could make it possible to identify precisely the types and frequencies of these sometimes asymptomatic, and probably underestimated, cardiac diseases.

The main questions it aims to answer are:

* To assess the incidence of AF and other cardiac arrhythmias and diseases occurring within 5 years after RT
* To evaluate absorbed doses in the heart and cardiac substructures (chambers, conduction nodes, coronaries, pulmonary veins) based on auto-segmentation models developped with deep learning algorithms
* To investigate whether the risk of AF and other cardiac arrhythmias and diseases is associated with cardiac irradiation characterized by these absorbed doses (dose-response relationship)

Participants will be included between 2023 and 2025, 5 years after their RT:

* Retrospective data collection will be based on a medical questionnaire designed to identify cardiac pathologies present prior to RT and those having occured in the past, between RT and 5 years post-RT.
* Cross-sectional data collection will be based on screening for cardiac pathologies using a connected watch worn for 1 month (silent AF screening) and a cardiology consultation (including ECG and echocardiography) to identify cardiac pathologies at 5 years post-RT possibly not identified in the retrospective data collection.

ELIGIBILITY:
Inclusion Criteria:

* Women treated surgically for primary cancer of the left or right breast and for whom adjuvant treatment is RT with irradiation of the breast or chest wall and possibly irradiation of lymph node chains,
* Adjuvant radiotherapy performed at Clinique Pasteur between 2018 and 2020,
* 5-year post-RT follow-up radiation oncologist consultation performed at Clinique Pasteur
* Age ≥ 65 years at the time of the 5-year post-RT follow-up consultation
* Own a smartphone and able to understand and use digital tools alone and/or with the help of a caregiver ;
* Patient having consented to connected follow-up,
* Be affiliated to a social security scheme or equivalent
* Be willing to participate in the study and have signed the consent form

Exclusion Criteria:

* History of cancer before breast cancer RT
* Recurrence of breast cancer or other cancer treated after breast cancer RT
* History of atrial fibrillation prior to breast cancer RT

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients treated with RT for breast cancer 5 years ago who come at radiotherapy service Clinique Pasteur for their last visit as part of the regular follow-up of patients by the radiation oncologist for 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of AF | 5 years
  AF previously diagnosed between RT and RT+5 years or silent AF incidentally diagnosed at 5-year post-RT screening

SECONDARY OUTCOMES:
Incidence of non AF cardiac arrhythmia | 5 years
  non AF arrhythmia previously diagnosed between RT and RT+5 years and/or incidentally diagnosed at 5-year post-RT screening
Incidence of other cardiac diseases | 5 years
  other cardiac diseases previously diagnosed between RT and RT+5 years and/or incidentally diagnosed at 5-year post-RT

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Jacob, PhD, Study Chair — Institut de Radioprotection et de Surete Nucleaire
Locations (1):
- Clinique Pasteur, Toulouse, France

REFERENCES:
- [Derived] Saint-Lary L, Pinel B, Panh L, Jimenez G, Geffrelot J, Kirova Y, Camilleri J, Broggio D, Bernier MO, Mandin C, Levy C, Boveda S, Thariat J, Jacob S. Screening and Risk Analysis of Atrial Fibrillation After Radiotherapy for Breast Cancer: Protocol for the Cross-Sectional Cohort Study "Watch Your Heart (WATCH)". JMIR Res Protoc. 2025 Jun 4;14:e67875. doi: 10.2196/67875. PMID 40466092